CLINICAL TRIAL: NCT04058145
Title: A Phase II Study of AMD3100 in Combination With Pembrolizumab in Head and Neck Squamous Cell Carcinoma Patients Who Have Progressed on Immune Checkpoint Blockade Therapy
Brief Title: AMD3100 Plus Pembrolizumab in Immune Checkpoint Blockade Refractory Head and Neck Squamous Cell Carcinoma
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Funding Withdrawn
Sponsor: Massachusetts General Hospital (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry); AperiSys, Inc (Unknown)
Responsible Party: Principal Investigator, Jong Chul Park, Principal Investigator, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 19-189
Record Dates: First submitted 2019-08-14; First posted 2019-08-15 (Actual); Last update posted 2020-09-07 (Actual); Status verified 2020-09

CONDITIONS: Head and Neck Cancer
Keywords: Head and Neck Cancer
MeSH Terms: conditions — Head and Neck Neoplasms | interventions — plerixafor; pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- Pembrolizumab+AMD3100 q3w (Experimental): * Pembrolizumab is administered intravenously on day 1 of each cycle
  * AMD3 100 is administered via injection subcutaneously on day 1 of each cycle
  Interventions: Drug: AMD3100; Drug: Pembrolizumab
- Pembrolizumab+AMD3100 weekly (Experimental): * Pembrolizumab is administered intravenously on day 1 of each cycle
  * AMD3 100 is administered via injection subcutaneously on a weekly basis
  Interventions: Drug: AMD3100; Drug: Pembrolizumab
- Pembrolizumab+AMD3100 (Experimental): * Pembrolizumab is administered intravenously
  * AMD3 100 is administered via injection subcutaneously
  Interventions: Drug: AMD3100; Drug: Pembrolizumab

INTERVENTIONS:
Drug: AMD3100 — AMD3100 is a drug that inhibits a chemokine CXCR4 which promotes cancer cell growth, spread, and survival and controls immune cell trafficking. Inhibiting CXCR4 expels the immune-suppressive cells out of the tumor and attract the cancer-killing immune cells into the tumor environment so that the body's immune system may be able to better attack the cancer cells.
  Other Names: Plerixafor
Drug: Pembrolizumab — Pembrolizumab is thought to block a receptor called PD-1. This receptor usually acts as a "brake" to prevent the body's immune system from attacking cancer cells. The antibody "removes the brake" to allow parts of the body's immune system (usually T cells) to attack the tumor.
  Other Names: Keytruda

SUMMARY:
This research is studying the safety and effectiveness of AMD3100 and pembrolizumab in participants with metastatic head and neck squamous cell carcinoma.

DETAILED DESCRIPTION:
This research study is a Phase II clinical trial. Phase II clinical trials test the safety and effectiveness of an investigational drug to learn whether the drug combination works in treating a specific disease. "Investigational" means that the drug is being studied.

Because AMD3100 and Pembrolizumab have not been administered together to individuals before, there will be a Run-In phase prior to the beginning of Phase II. This Run-In Phase is designed to identify what dosing schedule is best for participants on this study. Participants will be participating in the Run-In Phase.

The U.S. Food and Drug Administration (FDA) has approved Pembrolizumab as a treatment option for this disease.

The FDA has not approved AMD3100 as a treatment option for this disease, however it has approved the drug for use in individuals who have recently had bone marrow transplants.

Pembrolizumab is thought to block a receptor called PD-1. This receptor usually acts as a "brake" to prevent the body's immune system from attacking cancer cells. The antibody "removes the brake" to allow parts of the body's immune system (usually T cells) to attack the tumor

AMD3100 is a drug that inhibits CXCR4, which is a biological mechanism called a chemokine. CXCR4 is over-expressed in cancer cells and promotes cancer cell growth, spread, and survival and controls immune cell trafficking. Researchers believe that inhibiting CXCR4 expels the immune-suppressive cells out of the tumor and attract the cancer-killing immune cells into the tumor environment so that the body's immune system may be able to better attack the cancer cells.

In this research study, the investigators are assessing the safety and effectiveness of AMD3100 and pembrolizumab in participants with aggressive head and neck squamous cell carcinoma.

ELIGIBILITY:
Inclusion Criteria:

* Have histologically or cytologically confirmed diagnosis of squamous cell carcinoma of the recurrent or metastatic head and neck. For oropharyngeal cancer, tumor HPV status must be known.
* Have measurable disease based on RECIST 1.1. Lesions situated in a previously irradiated area are considered measurable if progression has been demonstrated in such lesions
* Have progressed on or after immune checkpoint therapy (anti-PD-1 or anti-PD-L1, as a monotherapy or in combination with other agents). Anti-PD-1/PD-L1 immune checkpoint therapy does not have to be the most immediate prior therapy before the study enrollment.
* Have provided archival tumor tissue sample or newly obtained core or excisional biopsy of a tumor lesion not previously irradiated. Formalin-fixed, paraffin embedded (FFPE) tissue blocks are preferred to slides. If slides are to be submitted, 10-20 unstained slides are required. Newly obtained biopsies are preferred to archived tissue. At a minimum, 3 core biopsies will be obtained and 1 core will be formalin fixed and the other 2 cores will be flash frozen.
* Have a lesion that is accessible for biopsy for subjects in the Run-In phase. An exception can be granted for those patients who do not have a lesion that can be safely biopsied based upon review with the Principal Investigator. The tumor biopsy is optional in the Phase II portion of the study
* Be >18 years of age on the day of signing informed consent.
* ECOG performance status ≤ 1 (Karnofsky ≥70%, see Appendix A).
* Have normal organ and marrow function as defined below. Specimens must be collected within 28 days prior to study registration.

  * leukocytes ≥3,000/mcL
  * absolute neutrophil count ≥1,500/mcL
  * platelets ≥100,000/mcL
  * total bilirubin ≤1.5 ×ULN
  * AST(SGOT)/ALT(SGPT) ≤2.5 × institutional upper limit of normal
  * creatinine Within normal institutional limits, OR
  * creatinine clearance ≥60 mL/min/1.73 m2 for participants with creatinine levels above institutional normal.
* Ability to understand and the willingness to sign a written informed consent document.
* Male participants:

A male participant must agree to use a contraception as detailed in Appendix C of this protocol during the treatment period and for at least 120 days after the last dose of study treatment and refrain from donating sperm during this period.

-Female participants:

A female participant is eligible to participate if she is not pregnant (see Appendix C), not breastfeeding, and at least one of the following conditions applies:

* Not a woman of childbearing potential (WOCBP) as defined in Appendix C, OR
* A WOCBP who agrees to follow the contraceptive guidance in Appendix C during the treatment period and for at least 120 days plus 30 days (a menstruation cycle) after the last dose of study treatment.

Exclusion Criteria:

* Has received prior systemic anti-cancer therapy including investigational agents within 2 weeks prior to registration with the exception of receiving immune checkpoint blockade therapy.
* Participants must have recovered from all AEs due to previous therapies to ≤ Grade 1 or baseline. Participants with ≤ Grade 2 neuropathy may be eligible after discussion with PI.
* Has received prior radiotherapy within 2 weeks of first dose of study drug.
* Participants must have recovered from all radiation-related toxicities to ≤Grade 1 or baseline, not require corticosteroids, and not have had radiation pneumonitis. A 1-week washout is permitted for palliative radiation (≤2 weeks of radiotherapy) to non-CNS disease.
* Has received a live vaccine within 30 days prior to the first dose of study drug. Examples of live vaccines include, but are not limited to, the following: measles, mumps, rubella, varicella/zoster (chicken pox), yellow fever, rabies, Bacillus Calmette-Guérin (BCG), and typhoid vaccine. Seasonal influenza vaccines for injection are generally killed virus vaccines and are allowed; however, intranasal influenza vaccines (eg, FluMist®) are live attenuated vaccines and are not allowed.
* Is currently participating in or has participated in a study of an investigational agent or has used an investigational device within 2 weeks prior to the first dose of study drug. Note: Participants who have entered the follow-up phase of an investigational study may participate as long as it has been >2 weeks since the last dose of the previous investigational agent.
* Has a known diagnosis of immunodeficiency or is receiving chronic systemic steroid therapy (in dosing exceeding 10 mg daily of prednisone equivalent) or any other form of immunosuppressive therapy within 7 days prior to the first dose of study drug.
* Has a known additional malignancy that is progressing or has required active treatment within the past 3 years. Note: Participants with basal cell carcinoma of the skin, squamous cell carcinoma of the skin, or carcinoma in situ (e.g. breast carcinoma, cervical cancer in situ) that have undergone potentially curative therapy are not excluded.
* Has known active CNS metastases and/or carcinomatous meningitis. Participants with previously treated brain metastases may participate provided they are radiologically stable, i.e. without evidence of progression for at least 4 weeks by repeat imaging (note that the repeat imaging should be performed during study screening), clinically stable and without requirement of steroid treatment for at least 14 days prior to first dose of study treatment.
* Has severe hypersensitivity (≥Grade 3) to pembrolizumab, AMD3100, and/or any of its excipients.
* Has active autoimmune disease that has required systemic treatment in the past 2 years (i.e. with use of disease modifying agents, corticosteroids or immunosuppressive drugs). Replacement therapy (eg., thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) is not considered a form of systemic treatment.
* Has a history of (non-infectious) pneumonitis that required steroids or has current pneumonitis.
* Has an active infection requiring systemic therapy.
* Has a known history of Human Immunodeficiency Virus (HIV).
* No HIV testing is required unless mandated by local health authority.
* Has a known history of Hepatitis B (defined as Hepatitis B surface antigen [HBsAg] reactive) or known active Hepatitis C virus (defined as HCV RNA [qualitative] is detected) infection. Note: No testing for Hepatitis B and Hepatitis C is required unless mandated by local health authority.
* Has a known history of active TB (Bacillus Tuberculosis).
* Has a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the study, interfere with the subject's participation for the full duration of the study, or is not in the best interest of the subject to participate, in the opinion of the treating investigator.
* Has known uncontrolled psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial.
* Is pregnant or breastfeeding or expecting to conceive or father children within the projected duration of the study, starting with the screening visit through 120 days after the last dose of trial treatment.
* A WOCBP who has a positive serum pregnancy test within 72 hours prior to registration (see Appendix C). Note: In the event that 72 hours have elapsed between the screening pregnancy test and the first dose of study treatment, another pregnancy test (urine or serum) must be performed and must be negative in order for subject to start receiving study medication.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2019-09-30 (Estimated); Primary Completion 2019-10-11 (Actual); Study Completion 2019-10-11 (Actual)

PRIMARY OUTCOMES:
Number of Participants That Experience a Dose Limiting Toxicity | From the start of treatment up to 24 months, or until disease progression or intolerable toxicity, whichever occurs first
  A safety run in will be conducted with AMD3100 administered weekly or every three weeks, both in combination with pembrolizumab administered every three weeks. The number of participants that experience dose limiting toxicities will be reported for each arm.
Overall Response Rate | From the start of treatment up to 24 months, or until disease progression or intolerable toxicity, whichever occurs first
  Overall response rate will be evaluated using Response Evaluation Criteria in Solid Tumors (RECIST). A participant is considered to have achieved a response if the achieve either of the following:
  * Complete Response (CR): Disappearance of all target lesions. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to <10 mm
  * Partial Response (PR): At least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters

SECONDARY OUTCOMES:
Progression Free Survival | From the time of randomization until disease progression or death, up to approximately 5 years
  The duration of time from randomization until disease progression or death. Disease progression is assessed using RECIST criteria.
  Confirmed Progressive Disease(CPD): At least a 20% increase in the sum of diameters of target lesions, taking as reference the smallest sum on study (this includes the baseline sum if that is the smallest on study). In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 mm. (Note: the appearance of one or more new lesions is also considered progression). Disease progression must be confirmed on a subsequent scan.
Overall Survival | From the time of randomization until death, up to approximately 5 years
  The median duration of time from the time of randomization until death.
The Number of Participants With Treatment-Related Serious Adverse Events | From the start of treatment until 30 days after the end of treatment, up to 25 months
  Adverse events are assessed using the NCI Common Terminology Criteria for Adverse Events (CTCAE) version 5.0. A treatment-related adverse event is an adverse event deemed to be possibly, probably, or definitely related to study treatment by the investigator.
Duration of Response | From the time of first response until disease progression, up to 24 months
  Duration of response is measured from the time measurement criteria are met for CR or PR (whichever is first recorded) until the first date that recurrent or progressive disease is objectively documented (taking as reference for progressive disease the smallest measurements recorded since the treatment started, or death due to any cause. Participants without events reported are censored at the last disease evaluation).

CONTACTS AND LOCATIONS:
Overall Officials: Jong Chul Park, MD, Principal Investigator — Massachusetts General Hospital
Locations (2):
- United States (2):
  - Massachusetts General Hospital Cancer Center, Boston, Massachusetts
  - Dana Farber Cancer Institute, Boston, Massachusetts

IPD SHARING:
Plan to Share IPD: Yes
The Dana-Farber / Harvard Cancer Center encourages and supports the responsible and ethical sharing of data from clinical trials. De-identified participant data from the final research dataset used in the published manuscript may only be shared under the terms of a Data Use Agreement. Requests may be directed to: [contact information for Sponsor Investigator or designee]. The protocol and statistical analysis plan will be made available on Clinicaltrials.gov only as required by federal regulation or as a condition of awards and agreements supporting the research
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data can be shared no earlier than 1 year following the date of publication
Access Criteria: MGH - Contact the Partners Innovations team at http://www.partners.org/innovation
URL: http://www.partners.org/innovation